CLINICAL TRIAL: NCT03070613
Title: Investigating the Use of Fluorescent Lectins to Identify Dysplasia and Cancer During Endoscopy and Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, TREVOR MING-YEE YEUNG, Academic Clinical Lecturer, University of Oxford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R37106
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Polyp
Keywords: Colonoscopy; Fluorescence guided surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescent Lectin Application (Experimental): Fluorescein conjugated wisteria floribunda will be sprayed onto the colonic surface during colonoscopy or TEM surgery.
  Interventions: Drug: Fluorescent Lectin Application

INTERVENTIONS:
Drug: Fluorescent Lectin Application — Fluorescein conjugated wisteria floribunda (a lectin).

SUMMARY:
This is a feasibility study investigating the use of a fluorescently conjugated lectin to identify colorectal dysplasia and cancer during colonoscopy and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 years or above
* Participants undergoing endoscopic procedures including colonoscopy and flexible sigmoidoscopy or transanal endoscopic microsurgery (TEMS), including robotic assisted TEMS
* In the investigator's opinion, is able and willing to comply with all study requirements

Exclusion Criteria

* Participant who is unable to unwilling to give informed consent
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial. If there is an uncertainty regarding whether a woman could be pregnant, then they will be excluded from the study
* Participants with known egg allergies, ovalbumin allergy and soya allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-23 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Signal to background ratios of identified colonic lesions under white light and under fluorescence | During procedure
  This outcome measure compares the fluorescence signal of lesions identified during colonoscopy.
Number of dysplastic and cancerous lesions identified under white light and under fluorescence | During procedure
  Number of lesions identified under white light colonoscopy will be compared to the number of lesions identified under fluorescence.

SECONDARY OUTCOMES:
Number of dysplastic and cancerous lesions identified under white light and fluorescence in different subgroups | 12 months
  Assessment of subgroups including ulcerative colitis, lesions suspicious of sessile serrated adenomas / traditional serrated adenomas
Resection margin of of lesions undergoing TEMS resection under white light and under fluorescence. | 12 months
  Planned resection margins will be compared under white light and under fluorescence. R0/R1 resection rates will be assessed post operatively.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Thomas Barnes, Oxford, Oxfordshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed